CLINICAL TRIAL: NCT03564184
Title: Longitudinal Study of Music Therapy's Effectiveness for Premature Infants and Their Caregivers: International Randomized Trial
Brief Title: Longitudinal Study of Music Therapy's Effectiveness for Premature Infants and Their Caregivers
Acronym: LongSTEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NORCE Norwegian Research Centre AS (Other)
Collaborators: Haukeland University Hospital (Other); University Hospital, Akershus (Other); Oslo University Hospital (Other); Meir Medical Center (Other); Clinica de La Mujer (Other); University of Haifa (Other); University of Gdansk (Other); King's College London (Other); Universidad de Ciencias Empresariales y Sociales (Unknown); Szpital Miejski w Rudzie Śląskiej (Unknown); SONO - Centro de Musicoterapia (Unknown); Hospital Materno Infantil Ramón Sardá (Network); Hospital Fernandez (Other)
Responsible Party: Principal Investigator, Christian Gold, Research Professor, NORCE Norwegian Research Centre AS
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: RCN 273534
Record Dates: First submitted 2018-06-10; First posted 2018-06-20 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Preterm Birth
Keywords: Parent-infant bonding; Music therapy
MeSH Terms: conditions — Premature Birth | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: 2x2 factorial, multinational, single-blind trial
Who Masked: Outcomes Assessor
Masking Description: Data collectors (for self-reports) and assessors (for observational measures) will be trained in assessment procedures and blinded to participant allocation. This will be ensured by using assessors from a different ward and by asking participants not to reveal their treatment assignments. Success of blinding will be verified.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MT during and after NICU (Experimental): Consists of music therapy during NICU hospitalization, and music therapy after discharge from initial NICU hospitalization, along with standard care.
  Interventions: Behavioral: MT during NICU; Behavioral: MT after NICU; Other: Standard care
- MT during NICU (Experimental): Consists of music therapy during NICU hospitalization, along with standard care.
  Interventions: Behavioral: MT during NICU; Other: Standard care
- MT after NICU (Experimental): Consists of music therapy after discharge from initial NICU hospitalization, along with standard care.
  Interventions: Behavioral: MT after NICU; Other: Standard care
- No MT (Experimental): Consists of standard care.
  Interventions: Other: Standard care

INTERVENTIONS:
Behavioral: MT during NICU — Music therapy (MT) by trained music therapist, 3 times/week for 30-40 minutes/session during NICU hospitalization. Involves primary caregiver and infant in musical communication matched to infant post-menstrual age, family/cultural preferences, and infant readiness for stimulation. Music therapist assesses infant´s needs and behavior state, supports caregiver in using basic touch (e.g., hand lightly and statically on infant´s chest or back to perceive breathing pattern) and caregiver´s hummed/sung voice matched to infant behavioral responses, to promote infant state regulation and bonding. Music includes input from music therapist as needed, and multimodal aspects such as gentle dynamic touch when infant demonstrates readiness. MT may occur while infant is held in a static manner by caregiver or is resting in his/her isolette or basinet. MT may occur during skin-to-skin care, if such care is part of standard care.
  Arms: MT during NICU; MT during and after NICU
Behavioral: MT after NICU — Music therapy offered by trained music therapist, 7 times for approximately 45 minutes/session across first 6 months following discharge from initial NICU hospitalization. Sessions include infant and caregiver, and siblings, if desired, and occur at home or in municipal settings. MT after NICU consists of a consult-to-parent model with each session including a brief verbal check-in regarding infant´s progress, musical interactions with music therapist modelling musical engagement, discussion of current challenges and strategies for using musical interactions to address needs in areas such as infant self-regulation, parent/infant interaction, and challenges with bonding. Caregivers will demonstrate techniques discussed during session, and form a brief plan for use of musical interaction in the interim before next session. Sessions will be adapted to infant developmental level and ongoing needs.
  Arms: MT after NICU; MT during and after NICU
Other: Standard care — Includes necessary medical care and standard supportive interventions offered as part of care during hospitalization, and standard follow-up procedures post-hospitalization.

SUMMARY:
Background: Preterm birth has major medical, psychological and socio-economic consequences worldwide. A recent systematic review suggests positive effects of music therapy (MT) on physiological measures of preterm infants and maternal anxiety, but methodologically rigorous studies including long-term follow-up of infant and parental outcomes are missing. Drawing upon caregivers' inherent resources, this study emphasizes caregiver involvement in MT to promote attuned, developmentally-appropriate musical interactions that may be of mutual benefit to infant and parent. This study will determine whether MT, as delivered by a qualified music therapist during neonatal intensive care unit (NICU) hospitalization and/or in home/municipal settings following discharge, is superior to standard care in improving bonding between primary caregivers and preterm infants, parent well-being and infant development.

Methods: Design: International multi-center, assessor-blind, 2x2 factorial, pragmatic randomized controlled trial. A feasibility study has been completed; ethical approval for the main trial is pending. Participants: 250 preterm infants and their parents. Intervention: MT focusing on singing specifically tailored to infant responses, will be delivered during NICU and/or during a post-discharge 6-month period. Primary outcome: Changes in mother-infant bonding until 6 months corrected age (CA), as measured by the Postpartum Bonding Questionnaire. Secondary outcomes: Mother-infant bonding at discharge and over 12 months CA; child development over 24 months; and parental depression, anxiety, and stress, and infant re-hospitalization, all over 12 months.

Discussion: This study fills a gap by measuring the long-term impact of MT for preterm infants/caregivers, and of MT beyond the hospital context. Outcomes related to highly involving parents in MT will directly inform the development of clinical practice in Scandinavia and other contexts with similar social welfare practices. By incorporating family-centered care, continuity of care, user involvement, and cultural relevance, this study can potentially contribute to improved quality of care for premature infants and their parents worldwide.

ELIGIBILITY:
Inclusion Criteria (infants):

* born below 35 weeks gestational age
* determined by medical staff to have achieved sufficient medical stability to start MT
* likely to be hospitalized longer than 2 weeks from time of recruitment

Inclusion Criteria (parents):

* willing to engage in at least 2 of 3 MT sessions per week during NICU and/or in 5 of 7 MT post-discharge sessions, if randomized to receive MT
* live with reasonable commuting distance from the treating NICU
* sufficient understanding of the respective national language(s) to answer questionnaires and participate in MT

Exclusion Criteria (parents):

* documented mental illness or cognitive impairment that prevents them from being able to complete the study intervention or outcome assessments

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2018-08-25 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Bonding between primary caregiver and infant | 6 months
  Total score of the Postpartum Bonding Questionnaire (PBQ), a parent-rated screening instrument for disorders of the early mother-infant relationship consisting of 25 statements on a six-point Likert scale (each 0-5; sum score ranging from 0 to 125; high = problematic).

SECONDARY OUTCOMES:
Bonding between primary caregiver and infant | 12 months
  Total score of the Postpartum Bonding Questionnaire (PBQ), a parent-rated screening instrument for disorders of the early mother-infant relationship consisting of 25 statements on a six-point Likert scale (each 0-5; sum score ranging from 0 to 125; high = problematic).
Child development | 24 months
  Bayley Scales of Infant and Toddler Development, 3rd edition (Bayley-III), standardized with a population mean of 100 (SD 15), with higher scores indicating better development
Infant development | 12 months
  Ages and Stages Questionnaire, 3rd edition (ASQ-3), an age-specific parent-reported screening questionnaire consisting of 30 items, total sum score ranging from 0 to 300, with higher scores indicating better development.
Infant socio-emotional development | 12 months
  Ages and Stages Questionnaire Social-Emotional (ASQ:SE), a parent-completed questionnaire with 19 or 22 Likert-scaled items (each 0-5-10), plus additional items for whether an item is of concern to the parent (each 0-5), resulting in a score ranging from 0-285 or 0-300, at 6 and 12 months respectively. Lower scores indicate better socio-emotional development.
Re-hospitalization | 12 months
  Re-hospitalization excluding outpatient visits, based on electronic health records. This will be calculated as the time from initial discharge until first re-hospitalization.
Maternal depression | 12 months
  Edinburgh Postnatal Depression Scale (EPDS), a 10-item validated self-report instrument assessing mothers' postpartum depressive symptoms, excluding somatic symptoms of depression that are common in new mothers (such as loss of energy, feeling tired, changes in appetite and sexual drive). Sum scores can range from 0 to 30, with high scores indicating more depressive symptoms.
Parental anxiety | 12 months
  Generalized Anxiety Disorder Assessment (GAD-7), a self-report 7-item questionnaire serving as a screening tool and severity measure for generalized anxiety disorder. Sum scores can range from 0 to 21, with higher scores indicating higher anxiety.
Parental stress | 12 months
  Parental Stress Scale (PSS), a self-report 18-item questionnaire that assesses stress associated with parenting. Sum scores can range from 18 to 90, with higher scores indicating higher stress.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Gold, PhD, Study Chair — NORCE Norwegian Research Centre; Claire Ghetti, PhD, Principal Investigator — Grieg Academy, University of Bergen
Locations (10):
- Argentina (3):
  - Hospital Materno Infantil Ramón Sardá, Buenos Aires, Buenos Aires F.D.
  - Sanatorio Mater Dei, Buenos Aires, Buenos Aires F.D.
  - Hospital Fernandez, Buenos Aires
- Colombia (2):
  - Clinica de la Mujer, Bogotá
  - Fundación Santa Fe de Bogotá, Bogotá
- Meir Medical Center, Kfar Saba, Israel
- Norway (3):
  - Haukeland University Hospital, Barne-og ungdomsklinikken, Bergen, Hordaland
  - Akershus University Hospital, Oslo, Lørenskog
  - Oslo University Hospital, Rikshospitalet, Oslo
- Szpital Miejski w Rudzie Śląskiej, Ruda Śląska, Poland

IPD SHARING:
Plan to Share IPD: Yes
To promote transparency and applicability of trial results and to facilitate re- analysis by other researchers while also protecting anonymity, de-identified individual patient data will be made available through the Norwegian Centre for Research Data (NSD).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Bieleninik L, Ghetti C, Gold C. Music Therapy for Preterm Infants and Their Parents: A Meta-analysis. Pediatrics. 2016 Sep;138(3):e20160971. doi: 10.1542/peds.2016-0971. Epub 2016 Aug 25. PMID 27561729
- [Background] Ghetti C, Bieleninik L, Hysing M, Kvestad I, Assmus J, Romeo R, Ettenberger M, Arnon S, Vederhus BJ, Soderstrom Gaden T, Gold C. Longitudinal Study of music Therapy's Effectiveness for Premature infants and their caregivers (LongSTEP): protocol for an international randomised trial. BMJ Open. 2019 Sep 3;9(8):e025062. doi: 10.1136/bmjopen-2018-025062. PMID 31481362
- [Derived] Bieleninik L, Kvestad I, Gold C, Stordal AS, Assmus J, Arnon S, Elefant C, Ettenberger M, Gaden TS, Haar-Shamir D, Havardstun T, Lichtensztejn M, Mangersnes J, Wiborg AN, Vederhus BJ, Ghetti CM. Music Therapy in Infancy and Neurodevelopmental Outcomes in Preterm Children: A Secondary Analysis of the LongSTEP Randomized Clinical Trial. JAMA Netw Open. 2024 May 1;7(5):e2410721. doi: 10.1001/jamanetworkopen.2024.10721. PMID 38753331
- [Derived] Ettenberger M, Bieleninik L, Stordal AS, Ghetti C. The effect of paternal anxiety on mother-infant bonding in neonatal intensive care. BMC Pregnancy Childbirth. 2024 Jan 11;24(1):55. doi: 10.1186/s12884-023-06179-z. PMID 38212696
- [Derived] Ghetti CM, Gaden TS, Bieleninik L, Kvestad I, Assmus J, Stordal AS, Aristizabal Sanchez LF, Arnon S, Dulsrud J, Elefant C, Epstein S, Ettenberger M, Glosli H, Konieczna-Nowak L, Lichtensztejn M, Lindvall MW, Mangersnes J, Murcia Fernandez LD, Roed CJ, Saa G, Van Roy B, Vederhus BJ, Gold C. Effect of Music Therapy on Parent-Infant Bonding Among Infants Born Preterm: A Randomized Clinical Trial. JAMA Netw Open. 2023 May 1;6(5):e2315750. doi: 10.1001/jamanetworkopen.2023.15750. PMID 37234006
- [Derived] Gaden TS, Gold C, Assmus J, Kvestad I, Stordal AS, Bieleninik L, Ghetti C. Treatment fidelity in a pragmatic clinical trial of music therapy for premature infants and their parents: the LongSTEP study. Trials. 2023 Mar 3;24(1):160. doi: 10.1186/s13063-022-06971-w. PMID 36869392
- [Derived] Gaden TS, Ghetti C, Kvestad I, Bieleninik L, Stordal AS, Assmus J, Arnon S, Elefant C, Epstein S, Ettenberger M, Lichtensztejn M, Lindvall MW, Mangersnes J, Roed CJ, Vederhus BJ, Gold C. Short-term Music Therapy for Families With Preterm Infants: A Randomized Trial. Pediatrics. 2022 Feb 1;149(2):e2021052797. doi: 10.1542/peds.2021-052797. PMID 34988583
- See also: Project website — https://www.norceresearch.no/en/projects/longitudinal-study-of-music-therapys-effectiveness-for-premature-infants-and-their-caregivers-longstep-international-randomized-trial